CLINICAL TRIAL: NCT05650671
Title: Measurement of Multiphysical Fields at the Subject-sitting Interface
Acronym: MECMISA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Other Study IDs: 2022_RIPH_006_MECMISA
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Wheelchair Users
Keywords: Wheelchair; Pressure ulcers; Pressure measurement; Temperature measurement; Humidity measurement
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- "wheelchair user-seat" group: healthy subjects agreeing to participate in the study
  Interventions: Device: instrumented wheelchair

INTERVENTIONS:
Device: instrumented wheelchair — Measurements of pressure, temperature and humidity at the subject/cushion interface

SUMMARY:
With the population ageing and the increase in disabilities prevalence, demand for wheelchairs is increasing. Padding and shape of seat are important factors for comfort when sitting for long periods of time. Sustained mechanical loads induced by the seated stance can cause pressure ulcers in the ischial prominences. Temperature and humidity have also been shown to be important in the development of pressure ulcers.

DETAILED DESCRIPTION:
The aim of this research is to measure the pressure, temperature and relative humidity fields at the user-seat interface of a wheelchair.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* aged of 18 and more
* agreeing to participate in the study

Exclusion Criteria:

* under 18 years old
* pregnant women

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
pressure | Day 0
  Pressures at the user-seat interface of a wheelchair will be measured by non-invasive method using a pressure pad positioned directly on the cushion, under the seated subject. No contact with the skin will take place
temperature | Day 0
  Temperatures at the ischial tuberosities will be measured by a non-intrusive methods using sensors taped directly on the pants of the participants. No contact with the skin of the participants will take place
humidity | Day 0
  Humidity at the ischial tuberosities will be measured by a non-intrusive methods using sensors taped directly on the pants of the participants. No contact with the skin of the participants will take place